CLINICAL TRIAL: NCT03861559
Title: Onset of Action of Mometasone Furoate (SCH 32088) Nasal Spray 50 mcg/Spray vs Placebo in Seasonal Allergic Rhinitis (Study No. C93-184).
Brief Title: Onset of Action of Mometasone Furoate (MK-0887/SCH 032088) Nasal Spray Compared With Placebo in Seasonal Allergic Rhinitis (C93-184)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C93-184; C93-184 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mometasone furoate nasal spray (Experimental): Participants administered mometasone furoate nasal spray 200 mcg once daily (QD), as two 50 mcg sprays per nostril, for 14 consecutive days.
  Interventions: Drug: mometasone furoate nasal spray
- placebo nasal spray (Placebo Comparator): Participants administered placebo nasal spray QD, as two placebo sprays per nostril, for 14 consecutive days.
  Interventions: Drug: placebo nasal spray

INTERVENTIONS:
Drug: mometasone furoate nasal spray — intranasal administration
  Other Names: NASONEX®; MK-0887; SCH 032088
  Arms: mometasone furoate nasal spray
Drug: placebo nasal spray — intranasal administration
  Arms: placebo nasal spray

SUMMARY:
This study investigated the onset of symptom relief following initiation of treatment with mometasone furoate (MK-0887/SCH 032088) 200 mcg administered once daily compared with placebo for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Has a 2-year history of seasonal allergic rhinitis
* Has a positive skin test response to a local seasonal allergen (current, or performed in investigator's office within the past year)
* Is in good health and free of any unstable, clinically-significant disease, other than allergic rhinitis, that would interfere with the study schedule or evaluation of seasonal allergic rhinitis

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women of childbearing potential who are not using an acceptable form of birth control
* Has asthma that requires therapy with inhaled or systemic corticosteroids, cromolyn, or nedocromil
* Has significant renal, hepatic, neurologic, cardiovascular, hematologic, metabolic, cerebrovascular, respiratory, gastrointestinal, or other significant medical illness or disorder which, in the judgment of the investigator, could interfere with the study, or required treatment which might interfere with the study
* Is on immunotherapy with the exception of maintenance therapy
* Has a clinically significant upper respiratory or sinus infection
* Has used an investigational drug within the previous 30 days
* Has nasal structural abnormalities, including large nasal polyps and marked septal deviation, that significantly interfere with nasal air flow
* Has a history of multiple drug allergies or an allergy to antihistamines or corticoids
* Has dependence upon nasal, oral or ocular decongestants, or nasal topical antihistamines, in the opinion of the investigator
* Has rhinitis medicamentosa
* Is using of any chronic medication which could affect the course of seasonal allergic rhinitis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 1994-03-30 (Actual); Primary Completion 1994-06-27 (Actual); Study Completion 1994-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 201 participants were randomized into the study (101 mometasone furoate; 100 placebo).
Groups:
- Mometasone Furoate Nasal Spray: Participants administered mometasone furoate nasal spray 200 mcg QD, as two 50 mcg sprays per nostril, for 14 consecutive days.
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 101 | 100
Completed | 99 | 95
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Treatment failure | 0 | 2
Not completed — Noncompliance | 1 | 1
Not completed — Did not meet eligibility requirements | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all participants who started the study and received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (10.1) | 31.8 (10.9) | 31.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 41 | 49 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 88 | 88 | 176
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Onset of Nasal Symptom Relief as Assessed by Participant Diary Responses
Description: Time to onset of relief of nasal stuffiness/congestion, rhinorrhea, nasal itching, sneezing, itching/burning eyes, tearing/watering eyes, redness of eyes, and itching of ears or palate was assessed by the participant using diary response data in the morning and night for the first 3 days of treatment. The participants were asked to rate their relief on the following scale: 1=complete, 2=marked, 3=moderate, 4=slight, and 5=none. If a participant recorded a degree of relief that was at least moderate (3 or below), they answered the question, "When did you first experience noticeable relief?" and noted the date and time. The data were analyzed using a log ranked test and with a Kaplan-Meier estimate. Any participant who did not experience at least moderate relief by the end of 72 hours was considered censored at that time in the analysis. Time to onset of relief is presented in hours.
Time Frame: From the start of treatment until onset of symptom relief (up to Day 4)
Population: Included randomized participants with ≥1 valid post-baseline visit, had evaluable data for the endpoint, and experienced at least moderate relief by the end of 72 hours of treatment.
Measure: Median (Full Range); unit: Hours
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 76 | 49
Hours | 35.9 [0.5 to 72.0] | 72.0 [0.25 to 72.0]
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, Log Rank

2. Secondary Outcome: Change From Baseline (CFB) in the Total Nasal Symptom Score (TNSS) Averaged Over 15 Days of Treatment, as Assessed by Participant
Description: CFB, averaged over study days 1-15, was calculated for TNSS assessed by participants. Participants scored 4 symptoms (rhinorrhea; nasal stuffiness; nasal itching; sneezing) in diaries using the scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. A decrease in symptom severity is reflected by a negative CFB.
  Percent CFB was calculated as the difference between the baseline and 15-day average scores divided by baseline score multiplied by 100. Scores were recorded twice daily, in morning (AM) and night (PM). Average AM/PM scores were first calculated separately, then averaged together to compute the 15-day average score. If diary entries were missing, an average AM or PM score was not calculated. If neither average AM nor PM score was calculated, total 15-day average score was not calculated. Baseline score was an average of the three AM and three PM scores preceding treatment.
Time Frame: Baseline (3 days preceding treatment) through Day 15 (averaged over 15 days)
Population: All randomized participants who took ≥1 dose of study medication, had ≥1 baseline endpoint observation, had ≥1 post-baseline visit, and evaluable data for the endpoint being analyzed. Baseline data was missing for 1 participant in the mometasone furoate nasal spray group for this endpoint and the participant was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 98
Percent change | -39 (2.0) | -20 (25.8)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

3. Other Pre Specified Outcome: Baseline Total Nasal Symptom Score (TNSS) for Calculation of Change From Baseline Averaged Over 15 Days of Treatment as Assessed by Participant
Description: TNSS was assessed by participants who scored 4 symptoms (rhinorrhea; nasal stuffiness; nasal itching; sneezing) in diaries using the scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. Scores were recorded twice daily, in morning (AM) and night (PM). The baseline score was an average of the three AM and three PM scores preceding treatment.
Time Frame: Baseline (3 days preceding treatment)
Population: All randomized participants who took ≥1 dose of study medication and provided ≥1 baseline endpoint observation for the calculation of the CFB in TNSS averaged over 15 days. Baseline data was missing for 1 participant in the mometasone furoate nasal spray group for this endpoint and the participant was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 98
Score on a scale | 8.4 (1.9) | 8.6 (1.7)

4. Secondary Outcome: Change From Baseline (CFB) in the Total Nasal Symptom Score (TNSS) at Day 4 as Assessed by Investigator
Description: CFB on study Day 4 was calculated for TNSS assessed by investigator. TNSS was a composite of the following symptoms: rhinorrhea, nasal stuffiness, nasal itching, and sneezing scores. The investigator scored each symptom during study visit on study Day 4, on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 4 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 4
Population: All randomized participants who took ≥1 dose of study medication, had ≥1 baseline endpoint observation, had ≥1 post-baseline visit, and evaluable data for the endpoint being analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 95
Percent change | -34 (28.8) | -16 (29.8)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

5. Secondary Outcome: Change From Baseline (CFB) in the Total Nasal Symptom Score (TNSS) at Day 8 as Assessed by Investigator
Description: CFB on study Day 8 was calculated for TNSS assessed by investigator. TNSS was a composite of the following symptoms: rhinorrhea, nasal stuffiness, nasal itching, and sneezing scores. The investigator scored each symptom during study visit on study Day 8 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 8 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 94
Percent change | -44 (33.4) | -28 (34.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

6. Secondary Outcome: Change From Baseline (CFB) in the Total Nasal Symptom Score (TNSS) at Day 15 as Assessed by Investigator
Description: CFB at Day 15 was calculated for TNSS assessed by the investigator. TNSS was a composite of the following symptoms: rhinorrhea, nasal stuffiness, nasal itching, and sneezing scores. The investigator scored each symptom during study visit on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and endpoint scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms. Signs and symptoms data collected by the investigator for Day 15 were not evaluated because the data was missing from the case report forms. The final endpoint was calculated using the last valid visit for each participant.
Time Frame: Baseline (Day 1) and Final Endpoint (Up to Day 15). The final endpoint was calculated using the last valid visit for each participant due to missing data at Day 15.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 98
Percent change | -43 (33.8) | -27 (34.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

7. Other Pre Specified Outcome: Baseline Total Nasal Symptom Score (TNSS) for Calculation of Change From Baseline at Days 4, 8, and 15 Visits as Assessed by Investigator
Description: TNSS was assessed by the investigator who scored 4 symptoms (rhinorrhea; nasal stuffiness; nasal itching; sneezing) in diaries using the scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12 where a higher value indicated greater severity. The baseline score was taken at the baseline visit preceding treatment.
Time Frame: Baseline (Day 1)
Population: All randomized participants who took ≥1 dose of study medication and provided at least 1 baseline endpoint observation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 98
Score on a scale | 8.9 (1.4) | 8.9 (1.7)

8. Secondary Outcome: Change From Baseline (CFB) in Overall Disease Condition Score at Day 4 as Assessed by Investigator
Description: CFB on study Day 4 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the investigator. The investigator scored the overall condition of the participant during the study visit on study Day 4 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 4 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 95
Percent change | -22 (30) | -16 (32.5)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.14, ANOVA

9. Secondary Outcome: Change From Baseline (CFB) in Overall Disease Condition Score at Day 8 as Assessed by Investigator
Description: CFB on study Day 8 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the investigator. The investigator scored the overall condition of the participant during the study visit on study Day 8 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 8 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 95
Percent change | -34 (35.5) | -22 (33.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.02, ANOVA

10. Secondary Outcome: Change From Baseline in Overall Disease Condition Score at Day 15 as Assessed by Investigator
Description: CFB on study Day 15 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the investigator. The investigator scored the overall condition of the participant during the study visit on study Day 15 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 15 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms. Signs and symptoms data collected by the investigator for Day 15 were not evaluated because the data was missing from the case report forms. The final endpoint was calculated using the last valid visit for each participant.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 94
Percent change | -41 (31.8) | -18 (30.7)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

11. Other Pre Specified Outcome: Baseline Overall Disease Condition Score for Calculation of Change From Baseline at Days 4, 8, and 15 Visits as Assessed by Investigator
Description: The investigator scored the overall condition of seasonal allergic rhinitis for the participant during the study visits using the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. The baseline score was taken at the baseline visit preceding treatment.
Time Frame: Baseline (Day 1)
Population: All randomized participants who took ≥1 dose of study medication and provided at least 1 baseline endpoint observation
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 98
Score on a scale | 2.3 (0.5) | 2.3 (0.4)

12. Secondary Outcome: Change From Baseline (CFB) in Overall Disease Condition Score at Day 4 as Assessed by Participant
Description: CFB on study Day 4 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the participant. The participant scored their overall condition on study Day 4 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 4 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 94
Percent change | -24 (33.5) | -18 (33.5)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.15, ANOVA

13. Secondary Outcome: Change From Baseline (CFB) in Overall Disease Condition Score at Day 8 as Assessed by Participant
Description: CFB on study Day 8 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the participant. The participant scored their overall condition on study Day 8 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 8 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 95
Percent change | -36 (34.0) | -21 (38.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

14. Secondary Outcome: Change From Baseline (CFB) in Overall Disease Condition Score at Day 15 as Assessed by Participant
Description: CFB on study Day 15 was calculated for the overall condition of seasonal allergic rhinitis as assessed by the participant. The participant scored their overall condition on study Day 15 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. Percent CFB was calculated as the difference between the baseline and Day 15 scores divided by baseline score multiplied by 100. A negative percent CFB indicated a decrease in symptom severity and a positive percent CFB indicated a worsening of symptoms.
Time Frame: Baseline (Day 1) and Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 94
Percent change | -41 (34.5) | -21 (37.0)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

15. Other Pre Specified Outcome: Baseline Overall Disease Condition Score for Calculation of Change From Baseline at Days 4, 8, and 15 as Assessed by Participant
Description: The participant scored the overall condition of seasonal allergic rhinitis in a diary using the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity. The baseline score was recorded preceding treatment.
Time Frame: Baseline (Day 1)
Population: All randomized participants who took ≥1 dose of study medication and provided at least 1 baseline endpoint observation
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 98
Score on a scale | 2.4 (0.5) | 2.4 (0.5)

16. Secondary Outcome: Therapeutic Response to Treatment at Day 4 as Assessed by Investigator
Description: Mean therapeutic response to treatment was assessed by evaluating the participant's relief of nasal symptoms during study visit on study Day 4. Treatment response was evaluated by the investigator using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms.
Time Frame: Day 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 95
Score on a scale | 3.2 (1.0) | 3.8 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

17. Secondary Outcome: Therapeutic Response to Treatment at Day 8 as Assessed by Investigator
Description: Mean therapeutic response to treatment was assessed by evaluating the participant's relief of nasal symptoms during study visit on study Day 8. Treatment response was evaluated by the investigator using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms.
Time Frame: Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 95
Score on a scale | 2.9 (1.1) | 3.5 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

18. Secondary Outcome: Therapeutic Response to Treatment at Day 15 as Assessed by Investigator
Description: Mean therapeutic response to treatment was assessed by evaluating the participant's relief of nasal symptoms during study visit on study Day 15. Treatment response was evaluated by the investigator using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms. Signs and symptoms data collected by the investigator for Day 15 were not evaluated because the data was missing from the case report forms. The final endpoint was calculated using the last valid visit for each participant.
Time Frame: Final Endpoint (Up to Day 15). The final endpoint was calculated using the last valid visit for each participant due to missing data at Day 15.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 94
Score on a scale | 2.7 (1.1) | 3.7 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

19. Secondary Outcome: Therapeutic Response to Treatment at Day 4 as Assessed by Participant
Description: Mean therapeutic response to treatment was assessed by the participant using diary cards on Day 4. Treatment response was evaluated by the participant using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms.
Time Frame: Day 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 99 | 94
Score on a scale | 3.2 (1.0) | 3.8 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

20. Secondary Outcome: Therapeutic Response to Treatment at Day 8 as Assessed by Participant
Description: Mean therapeutic response to treatment was assessed by the participant using diary cards on Day 8. Treatment response was evaluated by the participant using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms.
Time Frame: Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 98 | 95
Score on a scale | 2.9 (1.2) | 3.6 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

21. Secondary Outcome: Therapeutic Response to Treatment at Day 15 as Assessed by Participant
Description: Mean therapeutic response to treatment was assessed by the participant using diary cards on Day 15. Treatment response was evaluated by the participant using a 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group with a lower score indicating a greater response to treatment and an improvement in nasal symptoms.
Time Frame: Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 94
Score on a scale | 2.8 (1.1) | 3.6 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) and up to 14 days after study completion/discontinuation for non-serious adverse events and up to an additional 30 days after study completion for serious adverse events (up to 45 days).
Description: All participants who received at least one dose of study treatment and had at least one post-baseline evaluation for safety.
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 14/101 | 13/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=101) | Placebo Nasal Spray (N=99)
Headache (Nervous system disorders) | 14 (19) | 13 (19)

LIMITATIONS AND CAVEATS:
Adverse Event Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 12.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator and his co-workers agree not to publish or publicly present any results of the study without the prior written consent and approval of the sponsor.